CLINICAL TRIAL: NCT01887652
Title: Individualization of Controlled Ovarian Stimulation Using Anti-mullerian Hormone as a Biomarker of Ovarian Response Maximizes the Beneficial Effects of Treatment and Minimizes Complications and Risks.
Brief Title: Individualization of Ovarian Stimulation Using AMH Maximizes the Benefits and Minimizes Complications and Risks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ANDROFERT - Clinica de Andrologia e Reproducao Humana (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANDRO-03-12
Record Dates: First submitted 2013-06-24; First posted 2013-06-27 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Infertility
Keywords: In Vitro Fertilization; ovulation induction; anti-mullerian hormone
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional ovarian stimulation (Active Comparator): women whose protocol of ovarian stimulation was based on age, ovarian size and previous treatment
  Interventions: Other: conventional ovarian stimulation
- individualized ovarian stimulation (Active Comparator): women whose protocol of ovarian stimulation was based on anti-mullerian hormone
  Interventions: Other: individualized ovarian stimulation

INTERVENTIONS:
Other: conventional ovarian stimulation — a protocol of ovarian stimulation with recombinant FSH with dose according to age, ovarian size and previous treatment. In patients alder than 35, recombinant LH was added to ovarian stimulation.
  Arms: conventional ovarian stimulation
Other: individualized ovarian stimulation — After defining cut-off points of anti-mullerian hormone, using a ROC analysis, to discriminate excessive (≥20 oocytes retrieved) and poor response (≤4 oocytes retrieved), a individualized protocol was defined.Mild stimulation using daily doses (112.5 to 150 IU) of recombinant FSH or recombinant FSH combined with recombinant LH supplementation (375 IU total daily dose) were given to patients identified as at risk of excessive and poor response.
  Arms: individualized ovarian stimulation

SUMMARY:
The purpose oh the study is to determine the usefulness of anti-Mullerian hormone (AMH) to identify women at risk of excessive and poor response in controlled ovarian stimulation (COS) for in vitro fertilization (IVF), and the clinical impact of applying individualized COS strategies in these subsets of patients.

DETAILED DESCRIPTION:
A group of 130 women undergoing conventional COS after pituitary down-regulation for IVF will be studied to determine the best cut-off points of AMH, using receiver operating characteristic (ROC) analysis, to discriminate excessive (≥20 oocytes retrieved) and poor response (≤4 oocytes retrieved). The inclusion criteria is any patient with indication of IVF treatment. Subsequently, a different group of 120 women (with the same criteria) will be assessed using AMH before starting COS, and treatment strategy will be individualized according to AMH results (iCOS). Mild stimulation using daily doses (112.5 to 150 IU) of recombinant follicle stimulation hormone (rec-hFSH) or rec-hFSH combined with recombinant luteinizing hormone (LH) supplementation (375 IU total daily dose) will be given to patients identified as at risk of excessive and poor response, respectively. It will evaluated: number of oocytes, clinical pregnancy rates (defined as fetal heartbeat on ultrasound performed 4 weeks after the transfer of embryos) and occurrence of Ovarian hyperstimulation syndrome). Outcomes will be compared between the groups who received conventional and iCOS using chi-square and Fisher exact tests.

ELIGIBILITY:
Inclusion Criteria:

* women with in vitro fertilization treatment indication

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
number of oocytes retrieved | 1 day (on the day of oocyte retrieval)
  number of oocyte retrieved classified as: poor response: ≤4 oocytes normal response: 5 - 19 oocytes excessive response: ≥20 oocytes

SECONDARY OUTCOMES:
clinical pregnancy rate | 4 weeks after embryo transfer
  presence of fetal heartbeat on transvaginal ultrasound
occurrence of ovarian hyperstimulation syndrome | 4 weeks after embryo transfer
  presence of hyperstimulation syndrome during follow up after oocyte retrieval
cancellation | on the 8th day of ovarian stimulation
  cancellation of the cycle because of no ovarian response (no follicles >14 mm during ovarian stimulation)

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio BF Leao, MD, Principal Investigator — ANDROFERT - Clinica de Andrologia e Reproducao Humana; Sandro C Esteves, PhD, Study Director — ANDROFERT - Clinica de Andrologia e Reproducao Humana; Fabiana Y Nakano, Study Chair — ANDROFERT - Clinica de Andrologia e Reproducao Humana
Locations (1):
- Androfert, Campinas, São Paulo, Brazil